CLINICAL TRIAL: NCT01081990
Title: The Short-term Use of Cyclobenzaprine in Patients Undergoing Vaginal Surgery
Brief Title: Use of Cyclobenzaprine After Vaginal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EH10-073
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — cyclobenzaprine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Pill (Placebo Comparator)
  Interventions: Drug: cyclobenzaprine
- Flexeril (Experimental)
  Interventions: Drug: cyclobenzaprine

INTERVENTIONS:
Drug: cyclobenzaprine — Cyclobenzaprine 5 mg TID for 7 days

SUMMARY:
The management of post-operative pain in patients after vaginal surgery provides many unforeseen challenges. Although vaginal surgery is considered a minimally invasive approach for the repair of pelvic floor prolapse and urinary incontinence, patients may still experience varying degrees of discomfort and post-operative pain. Narcotics, however, can introduce a host of problems in addition to the potential addictive properties of the medication. A vicious cycle ensues as patients seek better pain control at the expense of worsening constipation, but without adequate control of pain after surgery, voiding dysfunctions are often exaggerated.

Cyclobenzaprine (Flexeril®) in conjunction with NSAIDs has long been the basis for management of acute musculoskeletal injuries, but the practice of prescribing this centrally acting muscle relaxant for post-operative patients has also been successful in the management of pain.

An online search of medical databases revealed that there are currently no published retrospective or prospective studies determining the efficacy of cyclobenzaprine in post surgical patients in conjunction with traditional pain management. The investigators hypothesize among healthy patients undergoing elective vaginal surgery for pelvic organ prolapse, the short-term use of a muscle relaxant could reduce the spasticity of the pelvic floor muscle attributable to surgery and thereby reduce the use of narcotics. Consequently, the reduction of narcotics and the control of post-surgical pain may also hasten the return of normal urinary and defecatory function.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70 years old
* Undergoing vaginal surgery with apical or posterior repair requiring hospitalization
* Willingness to participate in the study
* Normal neurological exam
* English speaking

Exclusion Criteria:

* Contraindication to NSAIDs
* Allergy to hydrocodone, hydromorphone, or cyclobenzaprine
* Renal disease
* Use of any antidepressants including SSRI, SNRI, MAOI in the last 3 months
* Glaucoma
* Diabetes
* Hyperthyroidism
* Uncontrolled hypertension (>160/100 mm Hg)
* History of chronic narcotic use in the last 3 months
* History of pelvic pain

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-04; Primary Completion 2014-07 (Actual); Study Completion 2014-08-01 (Actual)

PRIMARY OUTCOMES:
Faces Pain scale | 2 weeks
Quantity of pain medications | 2 weeks

SECONDARY OUTCOMES:
Constipation scale | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Jirschele, DO, Principal Investigator — Endeavor Health
Locations (1):
- Evanston NorthShore University HealthSystem, Evanston, Illinois, United States